CLINICAL TRIAL: NCT07099196
Title: Evaluating the Potential of Virtual Reality in Alleviating Pain and Anxiety Among Thalassemia Patients During Intravenous Cannulation: A Crossover Clinical Trial
Brief Title: Impact of Virtual Reality on Pain and Anxiety During Intravenous Cannulation Procedures Among Thalassemia Patients in UAE.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Bin Rashid University of Medicine and Health Sciences (Other)
Responsible Party: Principal Investigator, Sameer Asim Khan, MD Student, Mohammed Bin Rashid University of Medicine and Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MBRU-IRB-2024-80
Record Dates: First submitted 2025-07-05; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Thalassemia, Beta; Thalassemia; Pain; Anxiety; Blood Disorder
Keywords: thalassemia; Beta thalassemia; Virtual Reality; UAE; Pain; Anxiety; Intravenous cannulation; virtual reality therapy; medical hypnosis; digital health
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Pain; Anxiety Disorders; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalassemia patients (Experimental): This arm acts as its own control, with participants receiving SOC for their first visit, and then receiving VR for their next 2 visits during their cannulation procedure.
  Interventions: Device: Headset-based Virtual Reality Simulation

INTERVENTIONS:
Device: Headset-based Virtual Reality Simulation — The device used was a HEALTHY-MIND© PICO G2 Virtual Reality headset, which is medically graded and suited for distraction and relaxation in clinical settings.
  Other Names: Medical Hypnosis; Relaxation Tool; virtual reality; therapeutic virtual reality

SUMMARY:
The goal of this trial is to evaluate the effects of therapeutic Virtual Reality (VR) on pain, anxiety, fatigue and boredom during intravenous (IV) cannulations in comparison to standard of care (SOC).The main question it aims to answer is whether VR can act as an adjuvant for the IV cannulation procedure and improve overall patient experience.

Questionnaires were completed after the intravenous cannulation procedure during visits 1, 2 and 3. The Visual Analogue Scale (VAS) was used to assess both primary (pain and anxiety) and secondary (fatigue and boredom) objectives, collecting self-reported data during the three visits.

Heart Rate (measured in beats per minute (BPM)) and Blood Pressure (measured in millimeters of mercury (mmHg)) were measured after each procedure

* Participants will come for their routine cannulation and be recruited if willing
* Participants carry out the SOC procedure and are asked to fill out the questionnaires after
* The procedure is carried out with VR at the next appointment after 3-4 weeks
* This is repeated in the next visit

DETAILED DESCRIPTION:
Patients were screened at the Dubai Thalassemia Center during routine consultations, where the investigator present explained the study's objectives to the patient.

After consulting the patients' medical records and ensuring that there were no exclusion criteria and that the inclusion criteria were met, the investigators introduced themselves to the patients and their families, offering them the chance to take part in the study.

The investigators then explained to patients that they were eligible for this study and described the study's aims. Written, signed consent was obtained from adult patients and guardians of minors with an informed consent form.

Additionally, patients aged <18 years were provided with an assent form with simplified information about the study. Investigators took the time to answer the patient's questions about the study's progress, expected results, and anticipated benefits.

No financial compensation was paid to participants in this study. Participation in this study had no financial consequences for the participant, nor on his/her health insurance, as this was part of the routine care and consultation for the patient.

Participants were free to withdraw from the study at any time during the procedure. In the event of withdrawal, the data collected up to that point was analyzed, so as not to compromise the value of the study. Regardless of withdrawal, the anonymity of all patient data was maintained.

Interventions Patients benefited from the standard of care during their first visit, then utilized the VR intervention during the cannulation in their second visit and finally, another VR session in the third.

We used therapeutic immersions curated by the France-based company Healthy Mind, with various environments, including elements of medical hypnosis and breathing exercises, tailored for use in invasive procedures.

For each patient, the overall duration of the study was 6-8 weeks to complete all three visits, considering the 3-4 week interval between their scheduled appointments at the thalassemia center.

It should be noted that appointments were postponed if the patient did not complete the routine cross-matching test prior to the intravenous cannulation procedure or did not show up for their appointments.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of thalassemia
* Thalassemia patients undergoing intravenous cannulation procedure
* Patients aged >7 years (male, female, adult, pediatrics, national and non-national) at the Dubai Thalassemia Center

Exclusion Criteria:

Pregnant or nursing women

* Patients of legal age but subject to legal protection measures or unable to express their consent
* Patients suffering from uncontrolled epilepsy
* Patients with visual or auditory disorders
* Patients suffering from claustrophobia or motion sickness
* Patients with face infections
* Patients with dissociative psychiatric pathologies and/or autism

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Assessment of Pain using the Visual Analogue Scale | During the length of the cannulation procedure/VR session (between 10-20 minutes), at each clinical visit. Participants were scheduled for their next clinical visit/cannulation procedure exactly 2-4 weeks later, based on cross-matching results.
  Self-reported data assessed using the Visual Analogue Scale (VAS) ranging from 0 to 10, 0 is equivalent to no pain and 10 indicates the worst possible pain.
Assessment of Anxiety using the Visual Analogue Scale | During the length of the cannulation procedure/VR session (between 10-20 minutes), at each clinical visit. Participants were scheduled for their next clinical visit/cannulation procedure exactly 2-4 weeks later, based on cross-matching results.
  Self-reported data assessed using the Visual Analogue Scale (VAS) ranging from 0 to 10, Zero is equivalent to no anxiety and 10 indicates the worst possible anxiety.

SECONDARY OUTCOMES:
Assessment of Fatigue using the Visual Analogue Scale | During the length of the cannulation procedure/VR session (between 10-20 minutes), at each clinical visit. Participants were scheduled for their next clinical visit/cannulation procedure exactly 2-4 weeks later, based on cross-matching results.
  Self-reported data assessed using the Visual Analogue Scale (VAS) ranging from 0 to 10, 0 is equivalent to no fatigue and 10 indicates the worst possible fatigue.
Assessment of Boredom using the Visual Analogue Scale | During the length of the cannulation procedure/VR session (between 10-20 minutes), at each clinical visit. Participants were scheduled for their next clinical visit/cannulation procedure exactly 2-4 weeks later, based on cross-matching results.
  Self-reported data assessed using the Visual Analogue Scale (VAS) ranging from 0 to 10, 0 is equivalent to no boredom and 10 indicates the worst possible boredom.
Assessment of Patient Satisfaction | During the length of the cannulation procedure/VR session (between 10-20 minutes), at each clinical visit. Participants were scheduled for their next clinical visit/cannulation procedure exactly 2-4 weeks later, based on cross-matching results.
  Self-reported data using a questionnaire assessing their overall satisfaction, asking specific questions using the virtual reality headset during their second visit. (breathing exercises, chosen environment, feeling of relaxation etc..). Scale ranges from 'Very Dissatisfied' - 'Dissatisfied' - 'Neutral' - 'Satisfied' - 'Very Satisfied' - 'I don't know'.
Blood Pressure (mmHg) | After the cannulation procedure, at each clinic visit. Participants were scheduled for their next clinical visit/cannulation procedure exactly 2-4 weeks later, based on cross-matching results.
  Patient's vital signs were taken after the cannulation procedure
Heart Rate (BPM) | After the cannulation procedure, at each clinic visit. Participants were scheduled for their next clinical visit/cannulation procedure exactly 2-4 weeks later, based on cross-matching results.
  Patient's vital signs were taken after the cannulation procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Dubai Thalassemia Center, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study results will be published in aggregate form only.

REFERENCES:
- [Background] McLenon J, Rogers MAM. The fear of needles: A systematic review and meta-analysis. J Adv Nurs. 2019 Jan;75(1):30-42. doi: 10.1111/jan.13818. Epub 2018 Sep 11. PMID 30109720
- [Background] Gerceker GO, Bektas M, Aydinok Y, Oren H, Ellidokuz H, Olgun N. The effect of virtual reality on pain, fear, and anxiety during access of a port with huber needle in pediatric hematology-oncology patients: Randomized controlled trial. Eur J Oncol Nurs. 2021 Feb;50:101886. doi: 10.1016/j.ejon.2020.101886. Epub 2020 Dec 1. PMID 33321461
- [Background] Pandis N, Chung B, Scherer RW, Elbourne D, Altman DG. CONSORT 2010 statement: extension checklist for reporting within person randomised trials. BMJ. 2017 Jun 30;357:j2835. doi: 10.1136/bmj.j2835. PMID 28667088
- [Background] Wong CL, Lui MMW, Choi KC. Effects of immersive virtual reality intervention on pain and anxiety among pediatric patients undergoing venipuncture: a study protocol for a randomized controlled trial. Trials. 2019 Jun 20;20(1):369. doi: 10.1186/s13063-019-3443-z. PMID 31221208
- [Background] Walther-Larsen S, Petersen T, Friis SM, Aagaard G, Drivenes B, Opstrup P. Immersive Virtual Reality for Pediatric Procedural Pain: A Randomized Clinical Trial. Hosp Pediatr. 2019 Jul;9(7):501-507. doi: 10.1542/hpeds.2018-0249. Epub 2019 Jun 3. PMID 31160472
- [Background] Deacon B, Abramowitz J. Anxiety sensitivity and its dimensions across the anxiety disorders. J Anxiety Disord. 2006;20(7):837-57. doi: 10.1016/j.janxdis.2006.01.003. Epub 2006 Feb 8. PMID 16466904
- [Background] Neugebauer V, Li W, Bird GC, Han JS. The amygdala and persistent pain. Neuroscientist. 2004 Jun;10(3):221-34. doi: 10.1177/1073858403261077. PMID 15155061
- [Background] Wiederhold BK, Gao K, Sulea C, Wiederhold MD. Virtual reality as a distraction technique in chronic pain patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):346-52. doi: 10.1089/cyber.2014.0207. PMID 24892196
- [Background] Gold JI, Kim SH, Kant AJ, Joseph MH, Rizzo AS. Effectiveness of virtual reality for pediatric pain distraction during i.v. placement. Cyberpsychol Behav. 2006 Apr;9(2):207-12. doi: 10.1089/cpb.2006.9.207. PMID 16640481
- [Background] Mosso Vazquez JL, Mosso Lara D, Mosso Lara JL, Miller I, Wiederhold MD, Wiederhold BK. Pain Distraction During Ambulatory Surgery: Virtual Reality and Mobile Devices. Cyberpsychol Behav Soc Netw. 2019 Jan;22(1):15-21. doi: 10.1089/cyber.2017.0714. Epub 2018 Sep 25. PMID 30256662
- [Background] Chan JJI, Yeam CT, Kee HM, Tan CW, Sultana R, Sia ATH, Sng BL. The use of pre-operative virtual reality to reduce anxiety in women undergoing gynecological surgeries: a prospective cohort study. BMC Anesthesiol. 2020 Oct 9;20(1):261. doi: 10.1186/s12871-020-01177-6. PMID 33036555
- [Background] Chan E, Hovenden M, Ramage E, Ling N, Pham JH, Rahim A, Lam C, Liu L, Foster S, Sambell R, Jeyachanthiran K, Crock C, Stock A, Hopper SM, Cohen S, Davidson A, Plummer K, Mills E, Craig SS, Deng G, Leong P. Virtual Reality for Pediatric Needle Procedural Pain: Two Randomized Clinical Trials. J Pediatr. 2019 Jun;209:160-167.e4. doi: 10.1016/j.jpeds.2019.02.034. Epub 2019 Apr 29. PMID 31047650
- [Background] Rutter CE, Dahlquist LM, Weiss KE. Sustained efficacy of virtual reality distraction. J Pain. 2009 Apr;10(4):391-7. doi: 10.1016/j.jpain.2008.09.016. Epub 2009 Feb 23. PMID 19231295
- [Background] Aykanat Girgin B, Gol I. Reducing Pain and Fear in Children During Venipuncture: A Randomized Controlled Study. Pain Manag Nurs. 2020 Jun;21(3):276-282. doi: 10.1016/j.pmn.2019.07.006. Epub 2019 Sep 26. PMID 31501078
- [Background] Kazak AE, Kassam-Adams N, Schneider S, Zelikovsky N, Alderfer MA, Rourke M. An integrative model of pediatric medical traumatic stress. J Pediatr Psychol. 2006 May;31(4):343-55. doi: 10.1093/jpepsy/jsj054. Epub 2005 Aug 10. PMID 16093522
- [Background] Scalone L, Mantovani LG, Krol M, Rofail D, Ravera S, Bisconte MG, Borgna-Pignatti C, Borsellino Z, Cianciulli P, Gallisai D, Prossomariti L, Stefano I, Cappellini MD. Costs, quality of life, treatment satisfaction and compliance in patients with beta-thalassemia major undergoing iron chelation therapy: the ITHACA study. Curr Med Res Opin. 2008 Jul;24(7):1905-17. doi: 10.1185/03007990802160834. Epub 2008 May 27. PMID 18507891
- [Background] Al-Gazali L, Ali BR. Mutations of a country: a mutation review of single gene disorders in the United Arab Emirates (UAE). Hum Mutat. 2010 May;31(5):505-20. doi: 10.1002/humu.21232. PMID 20437613
- [Background] Baysal E. Molecular basis of beta-thalassemia in the United Arab Emirates. Hemoglobin. 2011;35(5-6):581-8. doi: 10.3109/03630269.2011.634706. PMID 22074124
- [Background] Baysal E. Hemoglobinopathies in the United Arab Emirates. Hemoglobin. 2001 May;25(2):247-53. doi: 10.1081/hem-100104033. PMID 11480786

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT07099196/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form: For Adults (>18yr) - English (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT07099196/ICF_001.pdf
  • Informed Consent Form: Assent Form: For Children (<18yr) - English (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT07099196/ICF_002.pdf